Date: December 14, 2024

## PATIENT INFORMATION AND CONSENT LETTER FOR THEIR PARTICIPATION IN A MEDICAL RESEARCH

Title of the research: Biological evolution of HELLP syndrome.

Dear Madam

We would like to invite you to take part in a clinical research study. This information letter explains what this study consists of. Please take the time to read and understand this information, to think about your participation and to ask the doctor in charge of the study to explain anything you may not have understood.

I. Aim of the study:

Analyze the biological evolution of HELLP syndrome in time before and after delivery.

II. Anticipated benefits:

Identify the different profiles that may respond to different therapies

III. Study process:

Clinical and biological data will be collected anonymously from your medical records.

IV. Potential risks:

As this is a simple questionnaire to fill in, no adverse effects are expected, and it will in no way affect the quality of your care. Responses are anonymous and no financial participation is expected.

V. Confidentiality:

Any information about you collected during this work will be treated as confidential.

Only the people in charge of the study, and possibly the health authorities, will have access to these data. With the exception of these people, who will process the information in strict compliance with medical secrecy, your anonymity will be preserved. Publication of the study results will not include any individual results, in accordance with the laws governing the processing of nominative data for health research purposes. If you have any questions during your participation in this study, please contact the doctors in charge of the study.

You are free to accept or refuse to take part in this study. This will not affect the quality of care you receive. Thank you for taking the time to read this letter. If you agree to participate in this research, we invite you to sign the enclosed consent form.

## **Consent form**

| participate in the study on the biological evolution of HELLP syndr | ,, 0 |
|---|---|
| The objectives and modalities of the study have been clearly explaor Dr Nizar Amllah. | ined to me by Pr Meryem ESSAFTI |
| I have read and understood the information sheet provided to me | |
| I accept that the documents in my medical file relating to the stud<br>managers and, if necessary, to the health authorities. With the ex-<br>handle the information in strict compliance with medical secrecy, | ception of these persons, who will |
| I understand that my participation in the study is voluntary. | |
| I am free to accept or refuse to participate, and I am free to stop r<br>the study. This will not affect the quality of care I receive. | ny participation at any time during |
| My consent does not relieve the organizers of this study of their reguaranteed by law. | esponsibilities. I retain all my rights |
| After discussion and after all my questions have been answered, I part in the proposed research. | freely and voluntarily agree to take |
| Signature of the patient: | Signature of the investigator : |